CLINICAL TRIAL: NCT01985945
Title: A Randomized Study of the Effect of Yoga in Patients With Breast Cancer Receiving Radiation Therapy
Brief Title: Yoga for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UPCC 08113
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Women With Stage I or II Breast Cancer Undergoing Active Radiation Therapy
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga (Other)
  Interventions: Other: Yoga
- Without Yoga (No Intervention)

INTERVENTIONS:
Other: Yoga
  Arms: Yoga

SUMMARY:
The purpose of this study is to examine the use of Eischens yoga for 8 weeks in one cohort of 20 women with stage I and II breast cancer receiving radiation therapy treatment, while a second cohort of the same type of and number of patients who, instead of yoga will receive standard supportive therapy, Questionnaire measuring cancer-related quality of life (FACT-G instrument) and fatigue (Brief Fatique Inventory) will be given to patients at several points.

ELIGIBILITY:
Inclusion Criteria:

* Stage I and II breast cancer patients undergoing active radiation therapy
* Above the age of 18
* Must sign informed consent form
* Must speak English
* Only women are eligible

Exclusion Criteria:

* Patients with medical restrictions that may interfere with yoga participation per their physicians' decision
* Those who have smoked in the last 6 months because smoking can interfere with the breathing and relaxation techniques of yoga.
* Those who have regularly taken yoga in the last 6 months, because they would not come to the intervention with the same baseline as other participants.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-03; Primary Completion 2015-07 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Gary Freedman, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States